CLINICAL TRIAL: NCT01415466
Title: A Randomized, Open Label, Multiple-Dose, Cross-over Clinical Study to Investigate Pharmacokinetics and Drug-Drug Interaction Between Rosuvastatin and CS-866 in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Drug Interaction Study Between Rosuvastatin and CS-866 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Collaborators: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_DWJ1276001
Record Dates: First submitted 2011-08-09; First posted 2011-08-12 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
MeSH Terms: interventions — Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- R (Experimental): multiple dose of Rosuvastatin 20mg
  Interventions: Drug: Cresto
- O (Experimental): multiple dose of CS-866 40mg
  Interventions: Drug: Olmetec
- R+O (Experimental): multiple dose of the combination of Rosuvastatin 20mg and CS-866 40mg
  Interventions: Drug: Cresto, Olmetec

INTERVENTIONS:
Drug: Cresto — tablet, 20mg
  Arms: R
Drug: Olmetec — tablet, 40mg
  Arms: O
Drug: Cresto, Olmetec — tablet, 20mg and 40mg
  Arms: R+O

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics profile and drug-drug interaction between rosuvastatin and CS-866 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male volunteers aged 20 to 50 years
2. A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints

Exclusion Criteria:

1. A subject who had any allergic history to any drug.
2. A subject with sign or symptoms or previously diagnosed disease of liver, kidney, neurology, respiratory, endocrinology, hematology, cardiovascular, genitourinary, psychology, ophthalmic, dermatology and gastrointestinal function or other significant diseases
3. History or suspicion of current drug abuse
4. A subject who had received treatment with below listed drug within specified period prior to the first dose of study medication

   * Within 1 month: drug known CYP inducer or inhibitor
   * Within 2 weeks: Prescribed or herbal medicine
   * Within 1 weeks: OTC medicine
   * Within 2 days: Consumption of caffeine
5. A subject who had participated in any other clinical study within the last 2 weeks
6. A subject from whom over 400mL of blood was sampled(whole blood donation) within last 2 weeks or plasma/platelet donation within 1 month.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
AUCtau | Multiple blood samples will be collected for 72 hours after last dosing in each of the periods.((in case of CS-866, for 48 hours)
Css,max | Multiple blood samples will be collected for 72 hours after last dosing in each of the periods.(in case of CS-866, for 48 hours)

SECONDARY OUTCOMES:
AUCss,last | Multiple blood samples will be collected for 72 hours after last dosing in each of the periods. (in case of CS-866, for 48 hours)
AUCss,inf | Multiple blood samples will be collected for 72 hours after last dosing in each of the periods. (in case of CS-866, for 48 hours)
Css,min | Multiple blood samples will be collected for 72 hours after last dosing in each of the periods. (in case of CS-866, for 48 hours)
T1/2 | Multiple blood samples will be collected for 72 hours after last dosing in each of the periods. (in case of CS-866, for 48 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsoo Park, M.D., Ph.D., Principal Investigator — YONSEI UNIVERSITY HEALTH SYSTEM (YUHS)
Locations (1):
- Yonsei University Health System (Yuhs), Seoul, South Korea